CLINICAL TRIAL: NCT02208609
Title: Absorption of Zinc (Zn) From Traditional Maize Tortillas and Amaranth-enriched Tortillas by Toddlers in the Indigenous Post-Mayan Population
Brief Title: Zinc Bioavailability From Amaranth-enriched Maize Tortillas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: International Atomic Energy Agency (Other Government); Universidad Francisco Marroquín (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 13-0282
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Nutritional Deficiency
Keywords: Zinc Absorption; Maize; Amaranth; Guatemala; Stable isotopes of Zn
MeSH Terms: conditions — Malnutrition; Callosities | interventions — Amaranth Dye

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maize Tortillas with 20% Amaranth (Experimental): Children in this arm were fed maize tortillas fortified with 20% amaranth
  Interventions: Other: Day 1: Maize Tortillas with 20% Amaranth
- Maize Tortillas without 20% Amaranth (Experimental): Children in this arm were fed maize tortillas without amaranth
  Interventions: Other: Day 2 Maize Tortillas without 20% Amaranth

INTERVENTIONS:
Other: Day 1: Maize Tortillas with 20% Amaranth — Subjects received Maize tortillas with 20% Amaranth added.
  Arms: Maize Tortillas with 20% Amaranth
Other: Day 2 Maize Tortillas without 20% Amaranth — Maize tortillas without Amaranth.
  Arms: Maize Tortillas without 20% Amaranth

SUMMARY:
Young children in Guatemala are at risk for nutrient deficiencies due to plant-based diets and poor sanitation. Stunting, frequent diarrhea, and respiratory infections are common. Supplementation of Zn to children during diarrhea episodes has been shown to diminish duration and severity of illness. Poor Zn absorption due to high fiber and phytate in this diet might play a role in these processes. Supplementation of this micronutrient in the diet might be beneficial. The investigators will compare absorption of Zn from white maize tortillas enriched with 20% amaranth to traditional white corn tortillas in preschool children in Guatemala.

DETAILED DESCRIPTION:
This is a randomized cross-over study of zinc absorption in young children living in the Western Highlands of Guatemala. Absorption of zinc will be measured from maize tortillas and maize tortillas fortified with 20% amaranth as the major food staple which provides at least 70% energy and at least 90% zinc and phytate of the diet. Participants will be randomized as to which type of tortilla they receive on the first and second day. Fractional absorption of zinc (FAZ) from all meals in one day for one type of tortilla and one day for the other will be measured by extrinsic labeling with stable isotopes of zinc. FAZ will be measured by a dual isotope tracer ratio (DITR) technique based on ratio of urine enrichment of orally versus intravenously administered zinc stable isotopes. Measurement of total zinc in duplicate diets on test days allow for determination of quantities of this micronutrient absorbed.

ELIGIBILITY:
Inclusion Criteria:

* 2-3 years of age
* apparently healthy
* eats >2-3 tortillas at each meal of the day.

Exclusion Criteria:

* Chispitas or macrovital supplementation
* breastfeeding
* birth weight < 2,500 g
* birth defect affecting growth and development
* chronic infection
* twin or triplet
* sibling enrolled in study

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Zinc Absorption | 2 days
  Absorption of zinc will be compared in young children when fed the common maize tortilla and a tortilla fortified with 20 % amaranth.. Fractional absorption of zinc for a day will be measured by extrinsic labeling with stable isotopes of zinc. Fractional absorption of zinc will be measured by a dual isotope tracer ratio technique. Measurement of total zinc in duplicate diets on test day will allow determination of quantity of this micronutrient absorbed (mg/d).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hambidge, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States
- Universidad Francisco Marroquin, Guatemala City, Guatemala

IPD SHARING:
Plan to Share IPD: No